CLINICAL TRIAL: NCT07064538
Title: A Mixed-Methods Open-Label Trial Evaluating the Effects of Neuralli® MP on Self-Defined Outcomes in Adults With Autistic Traits
Brief Title: Effects of Neuralli® MP on Self-Defined Outcomes in Adults With Autistic Traits
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shu-I Wu, Attending Physician, Mackay Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25CT027be
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: ASD; Autism; Autistic Disorders Spectrum
Keywords: Autistic traits; ASD
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuralli® MP (Experimental)
  Interventions: Dietary Supplement: Neuralli® MP

INTERVENTIONS:
Dietary Supplement: Neuralli® MP — Neuralli® MP containing 60 billion CFU (administered as two capsules per day)

SUMMARY:
To evaluate the efficacy of Neuralli® MP in improving participant-defined outcomes in adults with autistic traits.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a common neurodevelopmental disorder characterized by pervasive difficulties since early childhood across reciprocal social communication and restricted, repetitive interests and behaviors. Although early ASD research focused primarily on children, there is increasing recognition that ASD is a lifelong neurodevelopmental disorder. However, although health and education services for children with ASD are relatively well established, service provision for adults with ASD is in its infancy. There is a lack of health services research for adults with ASD, including identification of comorbid health difficulties, rigorous treatment trials (pharmacological and psychological), development of new pharmacotherapies, investigation of transition and aging across the lifespan, and consideration of sex differences and the views of people with ASD. The health services research for adults with ASD is urgently warranted. In particular, research is required to better understand the needs of adults with ASD, including health, aging, service development, transition, treatment options across the lifespan, sex, and the views of people with ASD.

Lactiplantibacillus plantarum PS128 (PS128), showed ameliorative effects on depression- and anxiety-like behaviors in different mouse models. When administered to children with ASD, PS128 was shown to improve anxiety, rule-breaking behaviors, hyperactivity/impulsivity, social function, inflammation index, and autonomic function. PS128 supplementation has also been shown to improve depressive symptoms and sleep quality for adults with self-reported insomnia, as well as cortisol levels and anxiety. However, even for this well-studied probiotic, its specific effects on broader aspects of ASD, such as core symptoms, cognition, attention, and sleep have not been systematically investigated.

Therefore, this study is designed not only to examine the effects of Neuralli® MP (PS128) but, more importantly, to explore the wider health and support needs of adults with autistic traits. By doing so, this study aims to assess how PS128 may contribute to improving their overall quality of life and address a range of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 50 who exhibit autistic traits
* Those who have the willingness and ability to work but have not yet been able to enter a sheltered workshop at the Kanner Foundation
* The subjects, primary caregivers and institution staff are willing to participate in the study, and the primary caregivers and institution staff are willing to fill out the questionnaire and accept the interview

Exclusion Criteria:

* Those who have taken antibiotics or probiotic products in powder, capsule or tablet form within the past month are excluded.
* Participants currently receiving antibiotic treatment are also excluded.
* Individuals with a known allergy to dairy products.
* Individuals with immunodeficiency or compromised immune function.
* Individuals diagnosed with small intestinal bacterial overgrowth (SIBO)
* Ineligibility determined by PI, e.g. the individual starts any new medication or therapy, especially related to their autism, during this time.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | weekly from baseline to week 8
  GAS is a method that can be used as a means of measuring outcome data from different contexts set out on a 5-point scale of -2 to +2.
  It enables the data to be placed on a quantitative measurement scale thus tackling the problem of how to adequately identify and measure qualitative goal impact and attainment. This is very useful as it enables a linking of measures from the frontline to upper levels of an organization's management.
  This assessment will be conducted weekly to determine how early the effects of the intervention can be observed.

SECONDARY OUTCOMES:
The Autism Behavior Checklist-Taiwan (ABCT) | from baseline to week 4 and week 8
  The Checklist scale contains 47 items: 8 items pertaining to sensory (sensation and perception), 11 items to relating (social connection), 12 items pertaining to body and object use (motor activity and rigid object use), 8 items pertaining to language (communication and interaction), and 8 items pertaining to social and self-Help (adaptability and self-care). The scoring method gives 1 point for each "Yes" answer. The higher the score, the more severe the autistic behaviors. This scale has favorable content consistency, with a Cronbach α value between 0.75 and 0.87, retest reliability at 0.89. The content validity and reliability of the scale are satisfactory.
Parent Target Symptom Rating Visual Analogue Scale (PTSVAS) | from baseline to week 4 and week 8
  A 100mm horizontal scale will be used to evaluate the descriptions and ratings, with each 10mm segment representing one unit. The scale ranges from "very good" or "completely resolved" (0) to "worst" or "catastrophic worsening" (10), with 5 representing no change.
Quality of Life in Autism Questionnaire (QoLA) | from baseline to week 4 and week 8
  The "Quality of Life in Autism Questionnaire" (QoLA) is a scale specifically designed for parents or caregivers of children with autism, aiming to assess their quality of life. The questionnaire consists of two parts:
  Part A: Evaluates the overall sense of quality of life experienced by the parent or caregiver. This section includes various items such as: "I feel happy and content" and "I am satisfied with my social life." Part B: Assesses the impact of the child's autism symptoms or characteristics on the parent or caregiver. The items in this section aim to understand how the child's autistic traits affect family life and the parent's daily experiences.
  The full questionnaire contains 48 items and is designed to comprehensively evaluate both the quality of life of the parent or caregiver and the impact of the child's autism symptoms on them.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided